CLINICAL TRIAL: NCT01503619
Title: Genomics of Small Cell Lung Carcinoma
Brief Title: Studying Biomarkers in Tumor Tissue and Blood Samples From Patients With Small Cell Lung Cancer Registered on CALGB-140202
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-151111; CDR0000721552 (Registry Identifier: NCI Physician Data Query); NCI-2012-00104 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2012-01-03; First posted 2012-01-04 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Lung Cancer
Keywords: small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (biomarker analysis): DNA isolated from archived tumor tissue and blood samples are analyzed for genetic mutations and gene expression profiling using Illumina exome sequencing. Results are compared with transcriptome of tumors (or cell lines) with and without the specific mutation. Cell culture studies overexpressing or inhibiting the genes of interest are also performed in a mouse model to identified potential drivers of small cell lung cancer.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tumor tissue and blood samples from patients with small cell lung cancer registered on CALGB-140202.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify the major genetic alterations in human small cell lung cancer (SCLC) using next-generation sequencing and focusing on mutations in coding sequence.

Secondary

* To follow up with in-depth assessment of candidate oncogenes and tumor suppressor genes using gene expression analysis, cell culture systems, and murine models of SCLC.

OUTLINE: DNA isolated from archived tumor tissue and blood samples are analyzed for genetic mutations and gene expression profiling using Illumina exome sequencing. Results are compared with transcriptome of tumors (or cell lines) with and without the specific mutation. Cell culture studies overexpressing or inhibiting the genes of interest are also performed in a mouse model to identified potential drivers of small cell lung cancer.

ELIGIBILITY:
* Patients must have been registered to CALGB-140202 trial in which tumor material (frozen tissue and paired blood specimens) is available
* Institutional Review Board (IRB) review and approval at the institution where the laboratory work will be performed is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with small cell lung cancer enrolled on the Cancer and Leukemia Group B (CALGB) 140202 study
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Identification of genetic alterations in human SCLC (driver or passenger mutations) | Baseline

SECONDARY OUTCOMES:
Gene expression between samples with or without mutations | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: David MacPherson, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States